CLINICAL TRIAL: NCT04944368
Title: A Phase II, Randomized, Two-armed, Double-blind, Placebo-controlled Trial to Evaluate the Safety, Tolerability, and Immunogenicity of an Adjuvanted Recombinant SARS-CoV-2 Spike (S) Protein Subunit Vaccine Candidate (SpikoGen)
Brief Title: Phase II Clinical Trial of CinnaGen COVID-19 Vaccine (SpikoGen)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cinnagen (Industry)
Collaborators: Vaxine Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC.CIN.PT.II; IRCT20150303021315N23 (Registry Identifier: Iranian Registry of Clinical Trials)
Record Dates: First submitted 2021-06-19; First posted 2021-06-29 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-01

CONDITIONS: Covid19
Keywords: COVID-19; SARS-COV-2; Recombinant protein; Spike; Advax-SM; Advax; Vaccine; Adjuvant
MeSH Terms: conditions — COVID-19 | interventions — SARS-CoV-2 recombinant spike protein with delta inulin and CpG-ODN adjuvant vaccine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine candidate (Experimental)
  Interventions: Biological: SARS-CoV-2 recombinant spike protein + Advax-SM adjuvant
- Saline placebo (Placebo Comparator)
  Interventions: Biological: Saline placebo

INTERVENTIONS:
Biological: SARS-CoV-2 recombinant spike protein + Advax-SM adjuvant — SARS-CoV-2 recombinant spike protein (25 µg) with Advax-SM adjuvant (15 mg) in two doses with a 21-day interval administered with intramuscular injections in the non-dominant arm
  Other Names: SpikoGen
  Arms: Vaccine candidate
Biological: Saline placebo — 0.9% sodium chloride (1 mL) injection in two doses with a 21-day interval administered with intramuscular injections in the non-dominant arm
  Other Names: Normal saline
  Arms: Saline placebo

SUMMARY:
This is a phase II, randomized, two-armed, double-blind, placebo-controlled trial designed to evaluate the safety, tolerability, and immunogenicity of a candidate adjuvanted recombinant SARS-CoV-2 spike (S) protein subunit vaccine (SpikoGen) produced by CinnaGen Co. 400 adult individuals receive either SARS-CoV-2 recombinant spike protein (25 µg) with Advax-SM adjuvant (15 mg) or saline placebo in a 3:1 ratio. The injection is given in two doses with a 21-day interval in the deltoid muscle of the non-dominant arm. The randomization was stratified by age (<65 or ≥65) and health conditions of potential risk for severe COVID-19. Participants will be visited at two weeks and will be followed up for six months after the second dose of the study intervention.

Study hypotheses include:

1. The adjuvanted COVID-19 vaccine candidate is safe and tolerable in adult subjects.
2. The adjuvanted COVID-19 vaccine candidate induces strong immunogenicity against SARS-CoV-2 in adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years
* Willing and able to comply with all study requirements, including scheduled visits, interventions, and laboratory tests
* Healthy adults or adults in a stable medical condition, defined as not being hospitalized within 3 months prior to the screening visit
* Females must not be pregnant or breastfeeding

Exclusion Criteria:

* Subjects with signs of active SARS-COV-2 infection at the screening visit.
* Subjects with body temperature of 38 degrees Celsius or greater at the screening visit or within 72 hours prior to the screening visit.
* Subjects with a history of any progressive or severe neurological disorders, seizure, or Guillain-Barre syndrome.
* Subjects who receive immunosuppressive or cytotoxic medications.
* Female Subjects who are pregnant or breastfeeding or have planned to become pregnant during the study period.
* Subjects who have a history of severe allergic reactions (e.g., anaphylaxis) to the study vaccine, any components of the study interventions, or any pharmaceutical products.
* Subjects who have received any other investigational products within 30 days prior to the screening visit or intend to participate in any other clinical studies during the period of this study.
* Subjects who have been vaccinated with any vaccine or vaccine candidate against SARS-CoV-2.
* Subjects who have received any vaccines within 28 days prior to the screening visit or intend to receive any vaccines up to 14 days after the second dose of the study injection.
* Subjects who have any known bleeding disorders or, in the investigator's opinion, have any contraindications for an intramuscular injection.
* Subjects who have received any blood, plasma, or immunoglobulin products from 90 days prior to the screening visit or intend to receive during the study period.
* Subjects with any condition that may increase the risk of participating in the study or may interfere with the evaluation of the primary endpoints of the study in the investigator's opinion.
* Subjects who have donated ≥450 mL of blood or blood products within 28 days prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of solicited adverse events | For 7 days after each dose
  Injection site pain, erythema, swelling, and induration, axillary swelling or tenderness ipsilateral to the side of injection, fever (oral temperature), headache, fatigue, myalgia, arthralgia, nausea, vomiting, and chills, as reported by the study participants on electronic diaries, and as defined using system organ classes and preferred terms of the Medical Dictionary for Regulatory Activities (MedDRA)
Incidence of unsolicited adverse events | For 28 days after each dose
  As reported by the study participants on electronic diaries, and as defined using system organ classes and preferred terms of the Medical Dictionary for Regulatory Activities (MedDRA)
Percentage of participants with seroconversion for S1 binding IgG antibodies after the first injection | 21 days after the first dose (on the day of the second dose)
  As measured by ELISA
Percentage of participants with seroconversion for S1 binding IgG antibodies after the second injection | 14 days after the second dose
  As measured by ELISA
Change in geometric mean concentration (GMC) for S1 binding IgG antibodies from baseline to 21 days after the first injection | On the day of the first dose and 21 days after the first dose (on the day of the second dose)
  As measured by ELISA
Change in geometric mean concentration (GMC) for S1 binding IgG antibodies from baseline to 14 days after the second injection | On the day of the first dose and 14 days after the second dose
  As measured by ELISA

SECONDARY OUTCOMES:
Percentage of participants with seroconversion for SARS-CoV-2 neutralizing antibodies after the first injection | 21 days after the first dose (on the day of the second dose)
  As measured by ELISA (sVNT)
Percentage of participants with seroconversion for SARS-CoV-2 neutralizing antibodies after the first injection | 21 days after the first dose (on the day of the second dose)
  As measured by cVNT
Percentage of participants with seroconversion for SARS-CoV-2 neutralizing antibodies after the second injection | 14 days after the second dose
  As measured by ELISA (sVNT)
Percentage of participants with seroconversion for SARS-CoV-2 neutralizing antibodies after the second injection | 14 days after the second dose
  As measured by cVNT
Percentage of participants with seroconversion for receptor-binding domain (RBD) binding IgA antibodies after the first injection | 21 days after the first dose (on the day of the second dose)
  As measured by ELISA
Percentage of participants with seroconversion for receptor-binding domain (RBD) binding IgA antibodies after the second injection | 14 days after the second dose
  As measured by ELISA
Percentage of participants with seroconversion for S1 binding IgA antibodies after the first injection | 21 days after the first dose (on the day of the second dose)
  As measured by ELISA
Percentage of participants with seroconversion for S1 binding IgA antibodies after the second injection | 14 days after the second dose
  As measured by ELISA
Percentage of participants with seroconversion for receptor-binding domain (RBD) binding IgG antibodies after the first injection | 21 days after the first dose (on the day of the second dose)
  As measured by ELISA
Percentage of participants with seroconversion for receptor-binding domain (RBD) binding IgG antibodies after the second injection | 14 days after the second dose
  As measured by ELISA
Change in geometric mean concentration (GMC) for receptor-binding domain (RBD) binding IgG antibodies from baseline to 21 days after the first injection | On the day of the first dose and 21 days after the first dose (on the day of the second dose)
  As measured by ELISA
Change in geometric mean concentration (GMC) for receptor-binding domain (RBD) binding IgG antibodies from baseline to 14 days after the second injection | On the day of the first dose and 14 days after the second dose
  As measured by ELISA
Geometric mean fold rise (GMFR) for S1 binding IgG antibodies after the first injection | 21 days after the first dose (on the day of the second dose)
  As measured by ELISA
Geometric mean fold rise (GMFR) for S1 binding IgG antibodies after the second injection | 14 days after the second dose
  As measured by ELISA
Geometric mean fold rise (GMFR) for receptor-binding domain (RBD) binding IgG antibodies after the first injection | 21 days after the first dose (on the day of the second dose)
  As measured by ELISA
Geometric mean fold rise (GMFR) for receptor-binding domain (RBD) binding IgG antibodies after the second injection | 14 days after the second dose
  As measured by ELISA
Geometric mean fold rise (GMFR) for SARS-CoV-2 neutralizing antibodies after the first injection | 21 days after the first dose (on the day of the second dose)
  As measured by ELISA (sVNT)
Geometric mean fold rise (GMFR) for SARS-CoV-2 neutralizing antibodies after the second injection | 14 days after the second dose
  As measured by ELISA (sVNT)
Change in geometric mean concentration (GMC) for SARS-CoV-2 neutralizing antibodies from baseline to 21 days after the first injection | On the day of the first dose and 21 days after the first dose (on the day of the second dose)
  As measured by ELISA (sVNT)
Change in geometric mean concentration (GMC) for SARS-CoV-2 neutralizing antibodies from baseline to 14 days after the second injection | On the day of the first dose and 14 days after the second dose
  As measured by ELISA (sVNT)
Change in geometric mean concentration (GMC) for S1 binding IgA antibodies from baseline to 21 days after the first injection | On the day of the first dose and 21 days after the first dose (on the day of the second dose)
  As measured by ELISA
Change in geometric mean concentration (GMC) for S1 binding IgA antibodies from baseline to 14 days after the second injection | On the day of the first dose and 14 days after the second dose
  As measured by ELISA
Geometric mean fold rise (GMFR) for S1 binding IgA antibodies after the first injection | 21 days after the first dose (on the day of the second dose)
  As measured by ELISA
Geometric mean fold rise (GMFR) for S1 binding IgA antibodies after the second injection | 14 days after the second dose
  As measured by ELISA
Incidence of serious adverse events (SAEs) and suspected unexpected serious adverse reaction (SUSARs) | For 6 months after the second dose
  As defined using system organ classes and preferred terms of the Medical Dictionary for Regulatory Activities (MedDRA)
Change in T-cell proliferation responses from baseline to 21 days after the first injection | On the day of the first dose and 21 days after the first dose (on the day of the second dose)
  Evaluation of CD4+ and CD8+ T-cell proliferation responses as measured by flow cytometry
Change in T-cell proliferation responses from baseline to 14 days after the second injection | On the day of the first dose and 14 days after the second dose
  Evaluation of CD4+ and CD8+ T-cell proliferation responses as measured by flow cytometry
Change in T-cell IFN-γ secretion from baseline to 21 days after the first injection | On the day of the first dose and 21 days after the first dose (on the day of the second dose)
  As measured by IGRA
Change in T-cell IFN-γ secretion from baseline to 14 days after the second injection | On the day of the first dose and 14 days after the second dose
  As measured by IGRA

CONTACTS AND LOCATIONS:
Overall Officials: Payam Tabarsi, M.D., Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Espinas Palace Hotel, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tabarsi P, Anjidani N, Shahpari R, Mardani M, Sabzvari A, Yazdani B, Roshanzamir K, Bayatani B, Taheri A, Petrovsky N, Li L, Barati S. Safety and immunogenicity of SpikoGen(R), an Advax-CpG55.2-adjuvanted SARS-CoV-2 spike protein vaccine: a phase 2 randomized placebo-controlled trial in both seropositive and seronegative populations. Clin Microbiol Infect. 2022 Sep;28(9):1263-1271. doi: 10.1016/j.cmi.2022.04.004. Epub 2022 Apr 15. PMID 35436611